CLINICAL TRIAL: NCT05292248
Title: Confidently Navigating Financial Decisions and Enhancing Financial Wellbeing in Dementia Caregiving
Brief Title: CONFIDENCE Financial Education for Caregivers
Acronym: CONFIDENCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Collaborators: AARP Foundation (Other); University of Southern California (Other)
Responsible Party: Principal Investigator, Kylie Meyer, Assistant Professor, Case Western Reserve University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20210794HU
Record Dates: First submitted 2022-03-14; First posted 2022-03-23 (Actual); Results first posted 2024-08-23 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Caregiver Burden; Financial Stress; Dementia; Alzheimer Disease
Keywords: Out-of-pocket costs; Behavioral intervention; Hispanic; Latino; Self-Efficacy
MeSH Terms: conditions — Caregiver Burden; Financial Stress; Dementia; Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CONFIDENCE Education Intervention (Experimental): Participants will attend the 5-week CONFIDENCEProgram. This program will include attending 5 group-based sessions delivered by videoconference. Each session will last approximately 1.5 hours each and will cover topics such as how to budget, accessing community resources to displace the out-of-pocket costs of caregiving, asking for help, balancing employment and caregiving, and more.
  Interventions: Behavioral: Confidently Navigating Financial Decisions and Enhancing Financial Wellbeing in Dementia Caregiving

INTERVENTIONS:
Behavioral: Confidently Navigating Financial Decisions and Enhancing Financial Wellbeing in Dementia Caregiving — Multicomponent psychoeducational intervention focused on financial wellbeing

SUMMARY:
The purpose of this study is to determine how feasible it is to deliver an online course to reduce out-of-pocket costs of caregiving and reduce financial stress among Latino family caregivers to a family member living with dementia. The investigators hope that that the results of this study will help to reduce high these out-of-pocket costs and improve financial wellbeing for Latino family caregivers.

Caregivers will be asked to to participate in 3 online surveys, in addition to participating in 5, 1.5 hour group-based Zoom learning sessions.

ELIGIBILITY:
Inclusion Criteria:

* Caregiver to someone diagnosed by a physician with probably Alzheimer's disease or a related dementia at least 6 months ago
* Latino or Hispanic ethnicity
* At least 50 years of age of older
* Able to attend 5, 1.5 hour to 2 hour group-based lessons over 5 weeks
* No plans to place family member in a facility within the next 3 months

Exclusion Criteria:

* Unreliable access to email, a computer and internet access
* Does note speak and read English
* Previously participated in CONFIDENCE program

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2024-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kylie Meyer, PhD, Principal Investigator — Case Western Reserve University
Locations (1):
- Case Western Reserve University, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data will be made available to qualified investigators upon request to the PI.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available, upon request, within 1 year of the study close date or the first publication using research data described, whichever comes first.
Access Criteria: Access will be provided using .csv files for de-identified study data and PDF supporting documents, sent by email.

REFERENCES:
- [Background] Rainville C, Skufca L, Mehegan L. Family Caregiving and Out-of-Pocket Costs: 2016 Report: AARP; 2016. https://www.khi.org/assets/uploads/news/14680/family-caregiving-cost-survey-res-ltc.pdf
- [Background] Norvilitis JM, Szablicki PB, Wilson SD. Factors Influencing Levels of Credit-Card Debt in College Students. J of Applied Social Psychology 2003;33(5):935-47.
- [Background] Ritter PL, Sheth K, Stewart AL, Gallagher-Thompson D, Lorig K. Development and Evaluation of the Eight-Item Caregiver Self-Efficacy Scale (CSES-8). Gerontologist. 2022 Mar 28;62(3):e140-e149. doi: 10.1093/geront/gnaa174. PMID 33146727
- [Background] Shim S, Barber BL, Card NA, Xiao JJ, Serido J. Financial socialization of first-year college students: the roles of parents, work, and education. J Youth Adolesc. 2010 Dec;39(12):1457-70. doi: 10.1007/s10964-009-9432-x. Epub 2009 Jul 4. PMID 20938727
- [Background] Shapiro GK, Burchell BJ. Measuring financial anxiety. Journal of Neuroscience, Psychology, and Economics. 2012;5(2):92-103.
- [Background] Zauszniewski JA, Lai CY, Tithiphontumrong S. Development and testing of the Resourcefulness Scale for Older Adults. J Nurs Meas. 2006 Spring-Summer;14(1):57-68. doi: 10.1891/jnum.14.1.57. PMID 16764178
- [Derived] Meyer K, Mage SM, Gonzalez A, Zauszniewski JA, Rhodes S, Perales-Puchalt J, Wilber K, Song L, Puga F, Benton D. Lessons from a Pilot Study of a Culturally Tailored Financial Well-Being Intervention Among Latino Family Caregivers. J Appl Gerontol. 2025 Jun;44(6):938-948. doi: 10.1177/07334648241293524. Epub 2024 Oct 17. PMID 39420566

RESULTS

PARTICIPANT FLOW:
Groups:
- CONFIDENCE Education Intervention: Participants attended the 5-week CONFIDENCEProgram. This program involved attending 5 group-based sessions delivered by videoconference. Each session lasted approximately 1.5 hours each and covered topics such as how to budget, accessing community resources to displace the out-of-pocket costs of caregiving, asking for help, balancing employment and caregiving, and more.
  Confidently Navigating Financial Decisions and Enhancing Financial Wellbeing in Dementia Caregiving: Multicomponent psychoeducational intervention focused on financial wellbeing
Period: Overall Study
Arm/Group | CONFIDENCE Education Intervention
Started | 20
Completed Intervention | 18
Follow Up Survey | 14
Completed | 14
Not Completed | 6

BASELINE CHARACTERISTICS:
Arm/Group | CONFIDENCE Education Intervention
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.6 (6.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 12
  More than one race | 1
  Unknown or Not Reported | 7
Region of Enrollment [Number; unit: participants]
  United States | 20
Monthly out-of-pocket caregiving costs [Median (Inter-Quartile Range); unit: Dollars] — Population: The number of participants with baseline data on out-of-pocket costs of care is lower than those who completed the baseline survey because 4 participants who completed the baseline survey did not complete the daily spending surveys.
  Dollars
    number analyzed (Participants) | 16
    (all) | 3755 [2537 to 5794.77]
Psychological financial strain [Mean (Standard Deviation); unit: units on a scale] — The measure for psychological financial strain is from multiple scales. Items 1 to 14 ask about financial anxiety. Lastly, the investigators included the 1-item question that asks about financial worry ("I worry constantly about money". Participants are asked to indicate the extent to which each statement is true (Very true [3], Somewhat true[2], Somewhat untrue[1], and Complete untrue[0]). Scores are summed such that scores range from 0 to 45, where higher scores indicate higher levels of financial strain.
  units on a scale | 17.9 (11.0)
Caregiver Self-Efficacy [Mean (Standard Deviation); unit: units on a scale] — Measured using the Caregiver Self-Efficacy Scale. This 8-item scale asks about multiple domains of self-efficacy. It demonstrates high reliability (alpha=0.89) and good test-retest reliability (0.73). Participants rate the extent to which they are "Not confident at all" (1) to "Totally confident" (10). Scores range from 8 (lowest level of self-efficacy) to 80 (highest level of self-efficacy). The outcome measure will use the average change score from baseline scores. Positive scores indicate an increase in self-efficacy. Population: One participant had missing data on this measure.
  units on a scale
    number analyzed (Participants) | 19
    (all) | 40.6 (13.5)
Resourcefulness [Mean (Standard Deviation); unit: units on a scale] — Resourcefulness is measured using the 28-item Caregiver Resourcefulness Scale (alpha=0.85). Caregivers are asked the frequency at which they use different strategies to manage challenges, and may respond: Not at all like me (0), Pretty much not like me (1), A little bit not like me (2), A little bit like me (3), Pretty much like much like me (4), or Very much like me (5). Items are added together to create a total score. Scores range from 0 to 140, where higher scores indicate higher levels of resourcefulness. The outcome measure will use the average change score from baseline scores Population: Four participants had missing data on this measure.
  units on a scale
    number analyzed (Participants) | 16
    (all) | 82.7 (26.0)

OUTCOME MEASURES:

1. Primary Outcome: Monthly Out-of-pocket Caregiving Costs
Description: Monthly out-of-pocket costs of caregiving is based on the tool used by the AARP Public Policy Institute in their 2016 report on the out-of-pocket costs of caregiving. This measure combines caregiver recall of care costs in the previous month, collected at baseline, with 5 days of daily spending diaries. Daily surveys will be sent using an email with a survey link, and a text message reminder. Monthly costs include less-frequent, high-cost expenditures (e.g., mortgage payment), while daily costs include lower-cost items caregivers may pay for more frequently (e.g., groceries). Daily self-reports of spending will be averaged and multiplied by 6 to approximate the number of days in a month, and added to estimated monthly costs.
  Positive scores indicate increased out-of-pocket costs. The researchers advise against relying on this outcome. In this pilot study, we found that this measure has qualitatively different meanings for adult child and spousal caregivers.
Time Frame: Change in median costs from from baseline to 8 weeks post-intervention
Population: Although all 20 participants were asked to complete daily spending surveys used to calculuate monthly out-of-pocket caregiving costs, only 16 completed daily spendin surveys at baseline. Of these participants, 10 completed daily spending surveys at the 2-month follow-up time. However, one follow-up survey was removed from analyses since it was an extreme outlier (i.e., 16 times higher than next highest monthly cost calculated).
Measure: Median (Inter-Quartile Range); unit: Dollars
Arm/Group | CONFIDENCE Education Intervention
Number analyzed (Participants) | 9
Dollars | 480 [149 to 994]

2. Secondary Outcome: Psychological Financial Strain
Description: The measure for psychological financial strain is from multiple scales. Items 1 to 14 ask about financial anxiety. Lastly, the investigators included the 1-item question that asks about financial worry ("I worry constantly about money". Participants are asked to indicate the extent to which each statement is true (Very true [3], Somewhat true[2], Somewhat untrue[1], and Complete untrue[0]). Scores are summed such that scores range from 0 to 45, where higher scores indicate higher levels of financial strain.
Time Frame: Change from baseline to post-intervention (within 1 week); change from baseline to 8 weeks post-intervention
Population: In both the first follow up and second follow up survey, there were 6 missing cases. In addition, for item-level missingness on this scale contributes to missing data for 2 additional cases.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CONFIDENCE Education Intervention
Number analyzed (Participants) | 14
score on a scale
  Change from baseline to post-intervention: number analyzed (Participants) | 12
  Change from baseline to post-intervention | -4.6 (7.8)
  Change from baseline to 8 weeks post-intervention: number analyzed (Participants) | 12
  Change from baseline to 8 weeks post-intervention | -4.3 (5.1)

3. Secondary Outcome: Caregiver Self-efficacy
Description: Self-efficacy is measured using the Caregiver Self-Efficacy Scale. This 8-item scale asks about multiples domains of self-efficacy (e.g., managing behavioral symptoms, accessing respite, and controlling upsetting thoughts). It demonstrates high reliability (alpha=0.89) and good test-retest reliability (0.73). Participants rate the extent to which they are "Not confident at all" (1) to "Totally confident" (10). Scores range from 8 (lowest level of self-efficacy) to 80 (highest level of self-efficacy). The outcome measure will use the average change score from baseline scores. Positive scores indicate an increase in self-efficacy.
Time Frame: Change from baseline to post-intervention (within 1 week); change from baseline to 8 weeks post-intervention
Population: A participant had item-level missingness at baseline, such that baseline data is available for 19 participants. Six participants did not complete the first follow up and the second follow up survey. Another participant had missing item-level data in the first follow up survey, such that there are 7 missing cases for "Change from baseline to post-intervention" and 6 missing cases for "Change from baseline to 8 weeks post-intervention."
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CONFIDENCE Education Intervention
Number analyzed (Participants) | 19
score on a scale
  Change from baseline to post-intervention: number analyzed (Participants) | 13
  Change from baseline to post-intervention | 15.2 (8.5)
  Change from baseline to 8 weeks post-intervention: number analyzed (Participants) | 14
  Change from baseline to 8 weeks post-intervention | 15.6 (6.5)

4. Secondary Outcome: Caregiver Resourcefulness
Description: Resourcefulness is measured using the 28-item Caregiver Resourcefulness Scale (alpha=0.85). This scale has two factors: one focused on help-seeking and another on self-help. Caregivers are asked the frequency at which they use different strategies to manage challenges, and may respond: Not at all like me (0), Pretty much not like me (1), A little bit not like me (2), A little bit like me (3), Pretty much like much like me (4), or Very much like me (5). Items are added together to create a total score. Scores range from 0 to 140, where higher scores indicate higher levels of resourcefulness. The outcome measure will use the average change score from baseline scores
Time Frame: Change from baseline to post-intervention (within 1 week); change from baseline to 8 weeks post-intervention
Population: Six participants did not complete the first follow up and the second follow up survey. In addition, two other participants had missing item-level data in the first follow up survey and another 4 had missing item-level data on the second follow up survey, such that there are 8 missing cases for "Change from baseline to post-intervention" and 10 missing cases for "Change from baseline to 8 weeks post-intervention."
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CONFIDENCE Education Intervention
Number analyzed (Participants) | 16
score on a scale
  Change from baseline to post-intervention: number analyzed (Participants) | 12
  Change from baseline to post-intervention | 12.8 (10.6)
  Change from baseline to 8 weeks post-intervention: number analyzed (Participants) | 10
  Change from baseline to 8 weeks post-intervention | 9.2 (9.7)

ADVERSE EVENTS:
Time Frame: 1 year, 5 months
Description: This was a benign behavioral intervention. We did not anticipate any serious adverse events, including mortality.
Arm/Group | CONFIDENCE Education Intervention
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-08-24): https://cdn.clinicaltrials.gov/large-docs/48/NCT05292248/Prot_SAP_000.pdf
  • Informed Consent Form (2022-08-16): https://cdn.clinicaltrials.gov/large-docs/48/NCT05292248/ICF_001.pdf